CLINICAL TRIAL: NCT01668004
Title: Open-Label, Phase 4 Study, Investigating the Incidence of Extra-Articular Manifestations in Subjects With Ankylosing Spondylitis Treated With Golimumab; Protocol No. MK-8259-012
Brief Title: The Incidence of Extra-Articular Manifestations in Participants With Ankylosing Spondylitis Treated With Golimumab (MK-8259-012)
Acronym: GO-EASY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8259-012; 2012-002458-21 (EudraCT Number)
Record Dates: First submitted 2012-08-01; First posted 2012-08-17 (Estimated); Results first posted 2016-08-03 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — golimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GLM 50 mg (Experimental): GLM given subcutaneously at a dose of 50 mg once monthly for up to 12 months
  Interventions: Biological: Golimumab

INTERVENTIONS:
Biological: Golimumab — GLM 50 mg subcutaneously once monthly.
  Other Names: Simponi®

SUMMARY:
The objective of this study is to determine the difference in the annual incidence rate of uveitis attacks in participants with ankylosing spondylitis (AS) before start initial anti-TNF therapy and after treatment with golimumab (GLM).

DETAILED DESCRIPTION:
This is an open-label, history-controlled, multi-site study of GLM in participants with AS. For evaluation of the primary study outcome measure, participants will serve as their own control. The period before start of treatment with an anti-tumor necrosis factor (TNF) agent will serve as historical control for the incidence of extra-articular manifestations, with a review of the medical records done for the previous 1-year period.

Each participant will participate in the study for approximately 12 months from the time the participant signs the Informed Consent Form through the final contact. After screening, two to four weeks before study start, each participant will be receiving study treatment for approximately 12 months, depending on the response to GLM after 3 months. All participants will be followed for a minimum of 12 months, irrespective of the duration of GLM treatment.

ELIGIBILITY:
Inclusion Criteria:

* May not have been treated with GLM prior to study enrollment
* Must be able to provide retrospective data concerning extra-articular manifestations and episodes with a recall period of at least 12 months prior to anti-TNF use
* Must have definite AS according to the modified New York criteria in the Netherlands
* Must be candidate for treatment with anti-TNF agent according to the Assessment of SpondyloArthritis International Society (ASAS) consensus
* Must be able to adhere to dose and visit schedules

Exclusion Criteria:

* Any exclusion criteria stated in the Summary of Product Characteristics for golimumab
* Use of any investigational biological or chemical agents within 30 days or 2 half-lives (whichever is longest) of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2012-09-03 (Actual); Primary Completion 2015-04-30 (Actual); Study Completion 2015-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Background] van Bentum RE, Heslinga SC, Nurmohamed MT, Gerards AH, Griep EN, Koehorst CBJM, Kok MR, Schilder AM, Verhoef M, van der Horst-Bruinsma IE. Reduced Occurrence Rate of Acute Anterior Uveitis in Ankylosing Spondylitis Treated with Golimumab - The GO-EASY Study. J Rheumatol. 2019 Feb;46(2):153-159. doi: 10.3899/jrheum.180312. Epub 2018 Nov 1. PMID 30385705

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 104 participants were screened; 3 participants were screen failures who did not enroll.
Groups:
- GLM 50 mg: Golimumab (GLM) given subcutaneously at a dose of 50 mg once monthly for up to 12 months
Period: Overall Study
Arm/Group | GLM 50 mg
Started | 101
Treated | 101
Completed | 76
Not Completed | 25
Not completed — Adverse Event | 7
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 5
Not completed — Lack of Efficacy | 9
Not completed — Non-compliance with treatment | 2

BASELINE CHARACTERISTICS:
Arm/Group | GLM 50 mg
Number analyzed (Participants) | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 66
Time since diagnosis [Mean (Standard Deviation); unit: Years] | 10.8 (11.8)
Age at onset of disease [Mean (Standard Deviation); unit: Years] | 33.1 (11.8)
Height [Mean (Standard Deviation); unit: cm] | 175.82 (9.62)
Weight [Mean (Standard Deviation); unit: kg] | 82.63 (18.00)
Abdominal circumference [Mean (Standard Deviation); unit: cm] | 95.5 (15.5)

OUTCOME MEASURES:

1. Primary Outcome: Occurence Rate of Uveitis Attacks in Participants Before Anti-TNF/GLM Treatment and After the Start of GLM Treatment
Description: Uveitis is an extra-articular manifestation of ankylosing spondylitis (AS) involving inflammation of the eye. The occurrence rate (assessed as present/absent) of uveitis attacks was determined over two 1-year long periods regardless of whether the event started during the assessed year: 1) the historical observation period consisting of the year before initial anti-TNF treatment (for anti-TNF experienced participants) or prior to first GLM dose (for anti-TNF naïve participants); and 2) the GLM observation period consisting of the year after first GLM dose.
Time Frame: Twelve Months Prior to Enrollment to Study Month 12
Population: All participants who received at least 3 months of GLM in the study and at least 3 months of follow-up data available for analysis of the endpoint (occurence of uveitis).
Measure: Number; unit: Ratio
Groups:
- Before Initial Anti-TNF/GLM Treatment: Historical observation period: Retrospective record review over the 12 months prior to the initial anti-TNF treatment (anti-TNF experienced participants) or the first GLM dose (anti-TNF naïve participants).
- After GLM Treatment Start: GLM observation period: Prospective follow-up of participants given GLM subcutaneously at a dose of 50 mg once monthly for up to 12 months
Arm/Group | Before Initial Anti-TNF/GLM Treatment | After GLM Treatment Start
Number analyzed (Participants) | 93 | 93
Ratio | 0.08 | 0.08
Statistical Analysis 1: Comparison: Before Initial Anti-TNF/GLM Treatment vs After GLM Treatment Start; Treatment comparison of uveitis occurrence rate assessed 1 year before initial anti-TNF/GLM treatment and 1 year after start of GLM treatment. Number of subjects included in analysis: N=93; Test type: Superiority or Other; p = 1.0000, McNemar

2. Primary Outcome: Annual Incidence Rate of New Uveitis Attacks in Participants Before Anti-TNF/GLM Treatment and After the Start of GLM Treatment
Description: Uveitis is an extra-articular manifestation of AS involving inflammation of the eye. The annual incidence rate of new uveitis attacks was determined over two 1-year long periods: 1) the historical observation period consisting of the year before initial anti-TNF treatment (for anti-TNF experienced participants) or prior to first GLM dose (for anti-TNF naïve participants); and 2) the GLM observation period consisting of the year after first GLM dose. All participants were counted as contributing a full year of GLM exposure even if discontinuing early. Due to ongoing uveitis cases at time of period entry, participants did not have the same risk of new events during the one year periods. Participants with ongoing uveitis at start of GLM who had the adverse event for the entire treatment period were counted as having the 'new attack' before and no "new attack" after GLM treatment start.
Time Frame: Twelve Months Prior to Enrollment to Study Month 12
Population: All participants who received at least 3 months of GLM in the study and at least 3 months of follow-up data available for analysis of the endpoint (incidence of uveitis). One participant for whom the timing of uveitis events could not be determined was excluded from the analysis.
Measure: Number; unit: Events per 100 participant years
Arm/Group | Before Initial Anti-TNF/GLM Treatment | After GLM Treatment Start
Number analyzed (Participants) | 92 | 92
Events per 100 participant years | 9.8 | 2.2
Statistical Analysis 1: Comparison: Before Initial Anti-TNF/GLM Treatment vs After GLM Treatment Start; Treatment difference (expressed as ratio) in uveitis incidence rate assessed 1 year before initial anti-TNF/GLM treatment and 1 year after start of GLM treatment. Number of subjects included in analysis: N=92; Test type: Superiority or Other; p < 0.0001, Generalized estimating equation; Treatment Ratio = 4.50, 95% CI 2-sided [3.86 to 5.25]

3. Secondary Outcome: Annual Incidence Rate of New-Onset or Flares of Inflammatory Bowel Disease (IBD) and Psoriasis in Participants Before Anti-TNF/GLM Treatment and After the Start of GLM Treatment
Description: IBD (Crohn's disease or ulcerative colitis) and psoriaris are extra-articular manifestations of AS involving the intestinal tract and skin, respectively. The annual incidence rates of new-onset or flares of IBD and psoriasis were to be determined separately (i.e., for each condition) over two 1-year long periods: 1) the historical observation period consisting of the year before initial anti-TNF treatment (for anti-TNF experienced participants) or prior to first GLM dose (for anti-TNF naïve participants); and 2) the GLM observation period consisting of the year after first GLM dose.
Time Frame: Twelve Months Prior to Enrollment to Study Month 12
Population: The incidence rates for new onset or flares of IBD and psoriasis could not be evaluated due to limitations of the data collected; occurrence of flares was not collected (specifically, history of IBD and/or psoriasis could not be distinguished from flares of IBD and/or psoriasis) and, therefore, results could not be determined.
Arm/Group | Before Initial Anti-TNF/GLM Treatment | After GLM Treatment Start
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Percentage of Bath Ankylosing Spondylitis Disease Activity Index 50 (BASDAI 50) Responders Following Treatment With GLM
Description: The percentage of participants with a BASDAI 50 response (defined as a 50% improvement or as an absolute improvement of 2 points in their BASDAI physical function score) at three months was determined. The BASDAI consists of total of six visual analog scales (VAS): five VAS (0 to 10 cm; increasing severity) measuring severity of fatigue, spinal pain, peripheral joint pain or swelling, localized tenderness, and severity of morning stiffness and one VAS (0 to 10 cm; increasing duration up to 2 hours) measuring duration of morning stiffness. The morning stiffness scores are averaged and summed with the scores for the remaining four items resulting in a composite score (0-50); the final BASDAI score (0-10) is derived by dividing by 5.
Time Frame: Baseline (BL), Study Month 3
Population: All participants who received at least 3 months of GLM in the study and at least 3 months of follow-up data available for analysis of the endpoint (BASDAI 50).
Measure: Number; unit: Percentage of participants
Arm/Group | GLM 50 mg
Number analyzed (Participants) | 88
Percentage of participants | 33.0

5. Secondary Outcome: Percentage of Ankylosing Spondylitis Disease Activity Score (ASDAS) Responders Following Treatment With GLM
Description: The percentage of participants with ASDAS clinically important improvement (ASDAS-CII; ≥ 1.1 units) and major improvement (ASDAS-MI; ≥ 2.0 units) at 3 months were determined. The ASDAS incorporates three items from the BASDAI (spinal pain, duration of morning stiffness, and peripheral joint pain or swelling) each assessed on a VAS (0 to 10 cm; increasing severity) as well as patient global assessment of disease activity (VAS; 0 to 10 cm; increasing severity) and a laboratory measure of inflammation (CRP level [mg/L] or ESR [mm/hr]). ASDAS was calculated using the formula: 0.12*Spinal Pain + 0.06*Duration of Morning Stiffness + 0.11*Patient Global + 0.07*Peripheral Pain/Swelling + 0.58*ln(CRP (mg/L) +1). A decrease in ASDAS at 3 months relative to BL signifies an improvement in physical function; ASDAS-MI (≥ 2.0 units decrease from BL) signifies a comparatively greater improvement in physical function than ASDAS-CII (≥ 1.1 units decrease from BL).
Time Frame: BL, Study Month 3
Population: All participants who received at least 3 months of GLM in the study and at least 3 months of follow-up data available for analysis of the endpoint (ASDAS).
Measure: Number; unit: Percentage of participants
Arm/Group | GLM 50 mg
Number analyzed (Participants) | 84
Percentage of participants
  ASDAS-CII (≥ 1.1 units) | 40.5
  ASDAS-MI (≥ 2.0 units) | 19.0

ADVERSE EVENTS:
Time Frame: Up to one year
Description: All safety analyses were performed on the All Treated Set, defined as all patients who received at least one dose of golimumab in the study. Only safety data during the GLM period was collected.
Arm/Group | GLM 50 mg
Serious Adverse Events (participants affected / at risk) | 7/101
Other Adverse Events (participants affected / at risk) | 21/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GLM 50 mg (N=101)
Acute Coronary Syndrome (Cardiac disorders) | 1 (1)
Cardiac Failure (Cardiac disorders) | 1 (1)
Colitis Ulcerative (Gastrointestinal disorders) | 1 (1)
Large Intestinal Ulcer Haemorrhage (Gastrointestinal disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Fistula Repair (Surgical and medical procedures) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GLM 50 mg (N=101)
Nasopharyngitis (Infections and infestations) | 11 (12)
Headache (Nervous system disorders) | 13 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the study. The sponsor shall have the right to review and comment with respect to publications, abstracts, slides, and manuscripts and the right to review and comment on the data analysis and presentation with regard to proprietary information, accuracy of information, and regulatory compliance.